CLINICAL TRIAL: NCT07068516
Title: A Multicenter, Randomized, Double-blind, Phase III Clinical Trial of Tislelizumab Combined With Chemotherapy Versus Placebo Plus Chemotherapy as Perioperative Treatment for MHC Class II-positive Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Perioperative Tislelizumab Plus Chemotherapy Versus Chemotherapy Alone in MHC-II-Positive Gastric/GEJ Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiangdong Cheng (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Principal Investigator, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mountain-04
Record Dates: First submitted 2025-06-15; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer Stage
MeSH Terms: interventions — tislelizumab; XELOX

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Placebo Comparator): Received placebo combined with investigator's choice of chemotherapy (either SOX or CAPOX regimen
  Interventions: Drug: SOX or CAPOX regimen
- Chemotherapy and immunotherapy (Experimental): Received tislelizumab combined with investigator's choice of chemotherapy (SOX or CAPOX regimen
  Interventions: Drug: Tislelizumab; Drug: SOX or CAPOX regimen

INTERVENTIONS:
Drug: Tislelizumab — Received tislelizumab combined with investigator's choice of chemotherapy
  Arms: Chemotherapy and immunotherapy
Drug: SOX or CAPOX regimen — chemotherapy (SOX or CAPOX regimen)

SUMMARY:
Investigators has conducted a series of studies on patient selection for perioperative immunotherapy in locally advanced gastric cancer. Results from prospective single-arm trial (NCT05739045) demonstrated that 21.74% of patients achieved pathological complete response (pCR) after receiving neoadjuvant nivolumab combined with SOX regimen. Notably, investigators identified that the sensitive group exhibited upregulated MHC-II expression in malignant cells at baseline, with enriched pathways including interferon-gamma signaling and MHC class II antigen presentation. The pCR rate was significantly higher in MHC-II positive patients compared to MHC-II negative patients (36.84% vs 11.11%, P=0.038). Subsequent retrospective analyses and another prospective single-arm study focusing on MHC-II positive populations consistently showed superior short-term treatment outcomes with immunotherapy plus chemotherapy in this subgroup.

Building upon these preliminary findings from small-scale studies and considering current developments in the field, we are now initiating this multicenter, randomized, double-blind, placebo-controlled phase III clinical trial. The study aims to evaluate the efficacy and safety of tislelizumab combined with chemotherapy versus placebo plus chemotherapy as perioperative treatment for MHC-II positive patients with locally advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and signed informed consent form
* ≥18 years old
* Histologically confirmed gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma
* MHC-II immunohistochemistry (IHC) 2+/3+
* Locally advanced disease (cT3-4a, N+, M0) confirmed by CT and/or diagnostic laparoscopy (AJCC 8th edition)
* No previous anticancer therapy (surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.)
* Scheduled to undergo curative resection after neoadjuvant therapy
* Ability to swallow oral medication
* ECOG performance status 0-1
* Estimated survival ≥6 months
* Hematological (without transfusion/G-CSF support within 14 days):ANC ≥1.5×10⁹/, Platelets ≥80×10⁹/L, Hemoglobin ≥80 g/L. Hepatic/Renal: Total bilirubin <1.5×ULN, ALT/AST ≤2.5×ULN, Serum creatinine ≤1.5×ULN or CrCl >50 mL/min (calculated by Cockcroft-Gault formula: Male: CrCl = [(140-age) × weight (kg)] / (72 × serum Cr [mg/dL]), Female: CrCl = [(140-age) × weight (kg)] / (72 × serum Cr [mg/dL]) × 0.85.
* Contraception Requirements: Female participants of childbearing potential: Negative serum pregnancy test within 7 days before enrollment; agreement to use highly effective contraception during treatment and for 120 days after last dose. Female participants of childbearing potential: Negative serum pregnancy test within 7 days before enrollment; agreement to use highly effective contraception during treatment and for 120 days after last dose.

Exclusion Criteria:

* Tumors deemed unresectable due to disease extent, surgical contraindications, or patient refusal.
* Known microsatellite instability-high (MSI-H) or mismatch repair-deficient (dMMR) tumors.
* History of or concurrent other malignancies (except adequately treated non-melanoma skin cancer or carcinoma in situ).
* Chronic or clinically significant conditions that may compromise treatment tolerance (e.g., severe cardiac disease, uncontrolled hypertension, significant hepatic/renal dysfunction).
* History of gastrointestinal perforation, intra-abdominal abscess, or bowel obstruction within 3 months (or clinical/radiologic suspicion of obstruction).
* Presence of active ulcers, non-healing wounds, or fractures.
* Arterial/venous thrombosis within 6 months (e.g., stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism).
* Urinalysis showing ≥++ protein with confirmed 24-hour urine protein >1.0 g.
* Requiring systemic antibiotics, antivirals, or antifungals.
* Hepatitis B: HBsAg-positive with HBV DNA ≥500 IU/mL. Hepatitis C: HCV antibody-positive with HCV RNA above ULN.
* Congenital or acquired (e.g., HIV infection).
* Active autoimmune disease or history of autoimmune disease with relapse potential.
* Prior or planned organ/allogeneic bone marrow transplantation.
* Interstitial lung disease (ILD), history of steroid-treated ILD, active pneumonia on screening CT, or active tuberculosis.
* Current or recent use of immunosuppressants or systemic corticosteroids (except physiologic replacement doses).
* Received live attenuated vaccines within 28 days before treatment or requiring them during/within 60 days post-treatment.
* Known allergy to any study drug or excipients.
* Currently breastfeeding.
* Any condition that, per investigator judgment, may jeopardize patient safety or study completion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | Perioperative
  To compare the pathological complete response (pCR) rates between tislelizumab plus chemotherapy and placebo plus chemotherapy as perioperative therapy for MHC-II-positive locally advanced gastric or gastroesophageal junction adenocarcinoma .

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No